CLINICAL TRIAL: NCT05472298
Title: The Effectiveness of Self-Management Skills and Technology in Individuals Who Have Both Metabolic Syndrome in Community
Brief Title: Effectiveness of Self-Management Skills for Metabolic Syndrome Fatty Liver Disease Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-Hung Chang, Professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MOST 107-2314-B-255-006
Record Dates: First submitted 2022-07-19; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Metabolic Syndrome
Keywords: self-management intervention; metabolic syndrome; women
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): lifestyle modification, goal setting, coaching and peer support, problem-solving, and self-monitoring
  Interventions: Behavioral: self-management intervention
- control arm (No Intervention): education leaflet

INTERVENTIONS:
Behavioral: self-management intervention — lifestyle modification, goal setting, coaching and peer support, problem-solving
  Arms: intervention arm

SUMMARY:
The multidimensional self-management intervention program focusing on healthy dietary habit and exercise effectively prevents metabolic syndrome. Thus, the purpose of this study was to assess the efficacy of multidimensional self-management intervention program on metabolic syndrome subjects in Taiwan.

DETAILED DESCRIPTION:
The study is a 2-parallel groups' randomized controlled trial. Participants with metabolic syndrome (three or more risk factors - triglycerides (TG) >150 mg/dL, systolic blood pressure (SBP) ≥130 mm Hg, diastolic blood pressure (DBP) ≥85 mm Hg, or fasting blood glucose≥100 mg/dL; high-density lipoprotein cholesterol<50 mg/dL, or waist circumference ≥80 cm) are enrolled. The four community units are randomized to receive a lifestyle intervention (intervention arm) or an education leaflet (control arm). The parameters are obtained from physical examination and biochemical assessments by well-trained case manager at baseline and each follow visit (6th months and 18th months). All participants complete a structured questionnaire, including basic information, physical activity, and food-frequency.

ELIGIBILITY:
Inclusion Criteria:

* adult women with age ≥ 50 years
* low education, defined as having less than 6 years of education or being primary school graduates
* presence of metabolic syndrome
* community-dwelling
* no hearing and visual acuity difficulties

Exclusion Criteria:

* Unconscious
* Cognitive impairment or dementia

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — adult women with age ≥ 50 years, low education, defined as having less than 6 years of education or being primary school graduates
Enrollment: 137 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
metabolic syndrome | 6 month, and 18-month follow up
  changes in triglycerides, high-density lipoprotein cholesterol, systolic blood pressure, diastolic blood pressure, fasting blood glucose, waist circumference

SECONDARY OUTCOMES:
body weight | 6 months, and 18 months follow up
  weight in kilograms
BMI | 6 months, and 18 months follow up
  weight and height will be combined to report BMI in kg/m^2

OTHER OUTCOMES:
leisure-time physical activity | 6 months, and 18 months follow up
  moderate-vigorous leisure-time physical activity at least 150 minutes a week
dietary behaviors | 6 months, and 18 months follow up
  intake rate of whole grains, vegetables, fruits, proteins, dairy products, and nuts.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hung Chang, Ph. D, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Taoyuan, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No